CLINICAL TRIAL: NCT01388335
Title: The Effect of Enzastaurin on CYP2C9: Enzastaurin - S-Warfarin Drug Interaction Study in Patients With Cancer
Brief Title: A Drug Interaction Study to Assess the Effect of LY317615 on the Metabolic Pathway of Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 9763; H6Q-MC-JCAX (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-07-04; First posted 2011-07-06 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumor; Lymphoma, Malignant
MeSH Terms: conditions — Lymphoma | interventions — Warfarin; enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- warfarin + enzastaurin (Experimental): On Day 1 of Period 1, a single 5-milligram (mg) oral dose of warfarin will be given, followed by at least a 7-day washout.
  Period 2: 500 mg enzastaurin administered orally once daily for at least 19 consecutive days and 5 mg warfarin administered as a single oral dose on Day 15.
  Safety Extension: Participants are allowed to continue receiving enzastaurin alone until disease progression or other discontinuation criteria are met.
  Interventions: Drug: warfarin; Drug: enzastaurin

INTERVENTIONS:
Drug: warfarin — Administered orally
Drug: enzastaurin — Administered orally
  Other Names: LY317615

SUMMARY:
The purpose of this study is to assess the effect of enzastaurin (LY317615), on a protein (enzyme CYP2C9) which is involved in the metabolic pathway of warfarin in participants with solid tumors or lymphomas. Information about any side effects that may occur will also be collected. This is a drug interaction study so the treatment of the disease will not be the main purpose of the study.

This is a Phase 1, open label, fixed sequence, 2 period study conducted in participants with solid tumors or lymphomas. The duration of participation in this study will be up to approximately 38 days not including screening, after which participants will be allowed to continue receiving enzastaurin. There is no planned duration for the extension phase of this study; participants will be allowed to continue to receive enzastaurin until fulfilling one of the criteria for discontinuation, such as unacceptable toxicity or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent approved by Eli Lilly and Company (Lilly) and the ethical review board (ERB) governing the site
* Have a histologic or cytologic diagnosis of cancer (lymphoma or solid tumor), with clinical or radiologic evidence of locally advanced and/or metastatic disease for which no life-prolonging therapy exists (Note: participants with glioblastoma, known central nervous system (CNS) metastases and other hematologic malignancies [except lymphoma] are excluded from this study)
* Men or women with reproductive potential must use an approved contraceptive method, if appropriate, during and for 3 months after discontinuation of study treatment. All methods of contraception should meet the criteria of highly effective contraceptives(failure rate of <1% per year) such as implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or vasectomized partner. Women with childbearing potential must have a negative serum pregnancy test ≤3 days prior to the first dosing day in the study (Period 1, Day 1).
* Have a performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) scale and, in the investigator's opinion, are suitable for participation in the study
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, anticancer hormone therapy, or other investigational therapy for at least 30 days prior to study entry (6 weeks for mitomycin-C or nitrosoureas), and have recovered from the acute effects of therapy
* For participants with hormone refractory prostate cancer, the following exception is permitted:

  * Participants receiving luteinizing hormone-releasing hormone (LHRH) analogue therapy (leuprolide, goserelin, or triptorelin) prior to starting this study should have that therapy continued while on this study.
  * In addition, participants who have received nonsteroidal antiandrogen therapy in the form of bicalutamide should have discontinued therapy at least 6 weeks prior to study entry (4 weeks if on flutamide or nilutamide).
* Have adequate organ function including:

  * Bone Marrow Reserve: absolute neutrophil count (ANC) ≥1.5 x 10˄9/liter (L) prior to treatment, platelets ≥100 x 10˄9/L, and hemoglobin ≥10 grams/deciliter (g/dL). Participants may receive erythrocyte transfusions to achieve this hemoglobin level at the discretion of the investigator. Participants may be allowed erythropoietin of choice as per standard of care.
  * Hepatic: bilirubin within 1.5 times the upper limit of normal (ULN), and transaminases ≤2.5 times ULN or ≤5 times ULN when liver metastases are known.
  * Renal: serum creatinine ≤1.5 milligrams/deciliter (mg/dL).
* Electrolytes: Participants may be entered into the study, if the investigator's opinion is that any electrolyte disorders, including potassium <3.4 milliequivalent per liter (mEq/L), calcium <8.4 mg/dL, or magnesium <1.2 mEq/L, may be appropriately managed and stabilized by the time of the laboratory evaluation on the baseline day in Period 1. If electrolytes have not been stabilized during this time, the participant will be discontinued from the study.
* Coagulation: normal prothrombin time/INR (PT/INR) and activated partial thromboplastin time (aPTT)
* Have an estimated life expectancy, in the judgment of the investigator, which will permit the participant to complete the drug interaction phase and at least 1 cycle of the safety extension phase (if the participant were to take part in the safety extension)

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with an experimental agent for non-cancer indications that has not received regulatory approval for any indication
* Participants with glioblastoma, Central Nervous System (CNS) metastases, or hematologic malignancies other than lymphoma are excluded from this study.
* Serious concomitant systemic disorder, including active infection, incompatible with the study (at the discretion of the investigator)
* History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infections
* Cardiac: Have a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV. Participants with a QTcB prolongation >450/470 millisecond (msec) (males/females) and participants who have a congenital long-QT-syndrome in their own or family medical history should be excluded at the investigator's discretion. Participants with intraventricular conduction delays (for instance, right or left bundle branch blocks) should also be excluded.
* It is recommended that participants with baseline arrhythmias (persistent or paroxysmal ventricular or supraventricular arrhythmias, including atrial fibrillation [occasional premature atrial contractions [APCs] or premature ventricular contractions [PVCs] are acceptable] or bradycardia (heart rate <50) be excluded, at the investigator's discretion.
* Known family history of unexplained sudden death
* Personal history of unexplained syncope within the last year
* The use of concomitant medications that prolong the QT/QTc interval
* Participants with complete gastrectomy or other significant GI diseases that, in the investigator's opinion, may significantly impact drug absorption
* Participants on total parenteral nutrition (TPN)
* Inability to swallow tablets
* Women who are lactating
* Participants with known allergies to enzastaurin or warfarin
* Participants with warfarin-related skin necrosis
* Participants who are known cytochrome P450 (CYP) 2C9 poor or intermediate metabolizers
* Drugs that are known inhibitors or inducers of CYP3A are specifically excluded. Foods that are known inhibitors of CYP3A (for example, grapefruit or grapefruit juice or Seville oranges or Seville orange juice) are also specifically excluded during Period 1 and Period 2 of the study.
* Drugs with narrow therapeutic windows and that are also known substrates of CYP2C9, CYP2C8, CYP2C19, and CYP3A are excluded.
* Use of any known inducers or inhibitors of CYP2C9 within 30 days (or at least 5 half-lives, whichever is shorter) prior to enrollment. Drugs that are inhibitors or inducers of CYP2C9 are also excluded throughout Periods 1 and 2. Drugs that are known to increase the hypoprothrombinemic effect of warfarin are excluded prior to enrollment and throughout Periods 1 and 2.
* Use of other anticoagulants or antithrombolytics within 14 days prior to screening or during Periods 1 and 2
* Use of low-dose aspirin (or higher doses) within 14 days prior to screening and during Period 1 and 2 of the study (allowed during continued safety extension phase)
* Use of high-dose acetaminophen (paracetamol) within 14 days of Period 1 and during Period 1 and 2 of the study
* Participants who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) or participants unwilling to stop alcohol consumption for the duration of the drug interaction phase (Periods 1 and 2) of the study (1 unit = 12 ounces (oz) or 360 milliliters (mL) of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Use of drugs of abuse, as evidenced by history, and/or positive findings on urinary drug screening, unless prescribed by a physician (for example, narcotic pain medication)
* Failure for any reason to satisfy the investigator for adequate fitness to participate in the study
* Major surgery or lumbar puncture in the past 6 weeks
* Protein C (functional) activity or Protein S antigen concentration below the normal range
* Heme-positive stool
* Warfarin is contraindicated in the case of congenital galactosemia, malabsorption syndromes of glucose and galactose, or lactase deficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse

RESULTS

PARTICIPANT FLOW:
Groups:
- Warfarin + Enzastaurin: Period 1 Day 1 (of an 8-day period): 5 milligrams (mg) warfarin administered as a single oral dose. Period included at least a 7-day washout.
  Period 2 (19 up to 30 days): 500 mg enzastaurin administered orally once daily for at least 19 consecutive days and 5 mg warfarin administered as a single oral dose on Day 15.
  Safety Extension Period: Participants were allowed to continue receiving 500 mg enzastaurin orally once daily alone until disease progression or other discontinuation criteria were met.
  Participants were on study for up to a total of 8 months (Period 1, Period 2 and Safety Extension Period).
Period: Period 1
Arm/Group | Warfarin + Enzastaurin
Started | 13
Received at Least 1 Dose of Study Drug | 13
Completed | 12
Not Completed | 1
Not completed — Progressive Disease | 1
Period: Period 2
Arm/Group | Warfarin + Enzastaurin
Started | 12
Received at Least 1 Dose of Study Drug | 12
Completed | 9 (Only 6 participants who completed Period 2 entered Safety Extension.)
Not Completed | 3
Not completed — Progressive Disease | 2
Not completed — Sponsor Decision | 1
Period: Safety Extension
Arm/Group | Warfarin + Enzastaurin
Started | 7 (Six completed Period 2 and 1 participant who discontinued Period 2 entered Safety Extension.)
Completed | 0
Not Completed | 7
Not completed — Progressive Disease | 7

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Warfarin + Enzastaurin: Period 1 Day 1 (of an 8-day period): 5 milligram (mg) warfarin administered as a single oral dose. Period included at least a 7-day washout.
  Period 2 (19 up to 30 days): 500 mg enzastaurin administered orally once daily for at least 19 consecutive days and 5 mg warfarin administered as a single oral dose on Day 15.
  Safety Extension Period: Participants were allowed to continue receiving 500 mg enzastaurin orally once daily alone until disease progression or other discontinuation criteria were met.
  Participants were on study for up to a total of 8 months (Period 1, Period 2 and Safety Extension Period).
Arm/Group | Warfarin + Enzastaurin
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
Region of Enrollment [Count of Participants; unit: Participants]
  France | 13

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of S-Warfarin and R-Warfarin
Description: Cmax of S-Warfarin and R-Warfarin determined using Geometric Least Squares (LS) mean model that was estimated from a mixed-effects model with repeated measures (MMRM) that included treatment as a fixed effect (warfarin alone as reference, and warfarin with enzastaurin as test), participant as a random effect and random error term.
Time Frame: Period 1 Day 1 (8 days) and Period 2 (19 up to 30 days): Predose, up to 96 hours postdose
Population: All enrolled participants who were assigned to a treatment, received at least 1 dose of study treatment.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms/milliliter (ng/mL)
Groups:
- Warfarin: Period 1 Day 1 (of an 8-day period): 5 milligrams (mg) warfarin administered as a single oral dose. Period included at least a 7-day washout.
- Warfarin + Enzastaurin: Period 2 (19 up to 30 days): 500 mg enzastaurin administered orally once daily for at least 19 consecutive days and 5 mg warfarin administered as a single oral dose on Day 15.
Arm/Group | Warfarin | Warfarin + Enzastaurin
Number analyzed (Participants) | 13 | 10
nanograms/milliliter (ng/mL)
  S-Warfarin | 245 [201 to 299] | 198 [161 to 245]
  R-Warfarin | 253 [214 to 298] | 230 [194 to 273]
Statistical Analysis 1: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Ratio = 0.810, 90% CI 2-sided [0.691 to 0.950] — Ratio of Geometric LS mean is for S-warfarin
Statistical Analysis 2: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Ratio = 0.912, 90% CI 2-sided [0.815 to 1.02] — Ratio of Geometric LS mean is for R-warfarin

2. Primary Outcome: Pharmacokinetics: Time of Maximal Plasma Concentration (Tmax) of S-Warfarin and R-Warfarin
Time Frame: Period 1 Day 1 (8 days) and Period 2 (19 up to 30 days): Predose, up to 96 hours postdose
Population: All enrolled participants who were assigned to a treatment and received at least 1 dose of study treatment and had S-warfarin and R-warfarin tmax values.
Measure: Median (Full Range); unit: hours
Arm/Group | Warfarin | Warfarin + Enzastaurin
Number analyzed (Participants) | 10 | 10
hours
  S-Warfarin | 2.04 [0.50 to 6.00] | 4.50 [2.02 to 8.02]
  R-Warfarin | 3.00 [0.50 to 12.0] | 7.00 [3.00 to 23.7]
Statistical Analysis 1: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Median Difference (Final Values) = 1.98, 90% CI 2-sided [0.76 to 3.50] — Median Difference (Final Values) is for S-warfarin
Statistical Analysis 2: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Median Difference (Final Values) = 2.50, 90% CI 2-sided [-1.00 to 6.84] — Median Difference (Final Values) is for R-warfarin

3. Primary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity [AUC(0-∞)] of S-Warfarin and R-Warfarin
Description: AUC(0-∞) determined using Geometric Least Squares (LS) mean model that was estimated from a mixed-effects model with repeated measures (MMRM) that included treatment as a fixed effect (warfarin alone as reference, and warfarin with enzastaurin as test), participant as a random effect and random error term.
Time Frame: Period 1 Day 1 (8 days) and Period 2 (19 up to 30 days): Predose, up to 96 hours postdose
Population: All enrolled participants who were assigned to a treatment and received at least 1 dose of study treatment and had S-warfarin and R-warfarin AUC(0-∞) values.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms*hours/milliliter (ng*h/mL)
Arm/Group | Warfarin | Warfarin + Enzastaurin
Number analyzed (Participants) | 13 | 9
nanograms*hours/milliliter (ng*h/mL)
  S-Warfarin | 8422 [7112 to 9973] | 10754 [9003 to 12846]
  R-Warfarin | 19122 [16471 to 22200] | 24058 [20350 to 28441]
Statistical Analysis 1: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Ratio = 1.28, 90% CI 2-sided [1.14 to 1.44] — Ratio of Geometric LS mean is for S-warfarin
Statistical Analysis 2: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Ratio = 1.26, 90% CI 2-sided [1.08 to 1.47] — Ratio of Geometric LS mean is for R-warfarin

4. Secondary Outcome: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) at Steady State of Enzastaurin, Its Principle Metabolites and Total Analyte
Description: Cmax at steady state (Cmax,ss) of enzastaurin, the principle metabolite (LSN326020), and the total analytes (enzastaurin, LSN326020, LSN485912 and LSN2406799) when enzastaurin is administered alone and with warfarin.
Time Frame: Period 2 Days 14 and 15 (19 up to 30 days): Predose, up to 24 hours postdose
Population: All enrolled participants who were assigned to a treatment and received at least 1 dose of study treatment and had Cmax,ss values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles/liter (nmol/L)
Groups:
- Enzastaurin: Period 2 (19 up to 30 days): 500 milligrams (mg) enzastaurin administered orally once daily for at least 19 consecutive days. Participants were allowed to continue receiving enzastaurin for 30 days, then either entered the Safety Extension Phase and continued receiving enzastaurin (up to a total of 8 months following the first dose of study drug) until disease progression or discontinued.
- Enzastaurin + Warfarin: Period 2 (19 up to 30 days): 500 mg enzastaurin administered orally once daily for at least 19 consecutive days and 5 mg warfarin administered as a single oral dose on Day 15.
Arm/Group | Enzastaurin | Enzastaurin + Warfarin
Number analyzed (Participants) | 10 | 10
nanomoles/liter (nmol/L)
  Enzastaurin | 2170 (93.3) | 2730 (85.3)
  Metabolite LSN326020 | 769 (56.5) | 872 (51.8)
  Total Analytes | 3600 (82.1) | 4410 (74.3)

5. Secondary Outcome: Pharmacokinetics: Time of Maximal Plasma Concentration (Tmax) of Enzastaurin, Its Principle Metabolites and Total Analyte
Description: Tmax at steady state (tmax,ss) of enzastaurin, the principle metabolite (LSN326020), and the total analytes (enzastaurin, LSN326020, LSN485912 and LSN2406799) when enzastaurin is administered alone and with warfarin.
Time Frame: Period 2 Days 14 and 15 (19 up to 30 days): Predose, up to 24 hours postdose
Population: All enrolled participants who were assigned to a treatment and received at least 1 dose of study treatment who had enzastaurin, LSN326020 and total analyte tmax,ss values.
Measure: Median (Full Range); unit: hours
Arm/Group | Enzastaurin | Enzastaurin + Warfarin
Number analyzed (Participants) | 10 | 10
hours
  Enzastaurin | 4.00 [0.00 to 8.08] | 4.00 [0.00 to 8.02]
  LSN326020 | 6.10 [2.00 to 8.08] | 8.01 [3.92 to 24.00]
  Total Analytes | 4.04 [0.00 to 9.08] | 4.02 [2.00 to 24.00]

6. Secondary Outcome: Pharmacokinetics: Area Under Concentration-Time Curve Over a Dosing Interval at Steady State (AUCss) of Enzastaurin, Its Principle Metabolites and Total Analyte
Description: AUCss of enzastaurin, the principle metabolite (LSN326020), and the total analytes (enzastaurin, LSN326020, LSN485912 and LSN2406799) when enzastaurin is administered alone and with warfarin.
Time Frame: Period 2 Days 14 and 15 (19 up to 30 days): Predose, up to 24 hours postdose
Population: All enrolled participants who were assigned to a treatment and received at least 1 dose of study treatment who had enzastaurin, LSN326020 and total analyte AUC,ss values .
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour/liter (nmol*h/L)
Arm/Group | Enzastaurin | Enzastaurin + Warfarin
Number analyzed (Participants) | 10 | 10
nanomoles*hour/liter (nmol*h/L)
  Enzastaurin | 35200 (124) | 44100 (115)
  LSN326020 | 16300 (64.0) | 19000 (53.2)
  Total Analytes | 64800 (103) | 80500 (94.1)

7. Secondary Outcome: Pharmacokinetics: Average Concentration During a Dosing Interval Steady State (Cav,ss) of Enzastaurin, Its Principle Metabolites and Total Analyte
Description: Cav,ss of enzastaurin, the principle metabolite (LSN326020), and the total analytes (enzastaurin, LSN326020, LSN485912 and LSN2406799) when enzastaurin is administered alone and with warfarin.
Time Frame: Period 2 Days 14 and 15 (19 up to 30 days): Predose, up to 24 hours post dose
Population: All enrolled participants who were assigned to a treatment and received at least 1 dose of study treatment who had enzastaurin, LSN326020 and total analyte Cav,ss values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | Enzastaurin | Enzastaurin + Warfarin
Number analyzed (Participants) | 10 | 10
nanomole/liter (nmol/L)
  Enzastaurin | 1470 (124) | 1840 (115)
  LSN326020 | 680 (64.0) | 790 (53.2)
  Total Analytes | 2700 (103) | 3350 (94.1)

8. Secondary Outcome: Pharmacodynamics: Maximum International Normalised Ratio (INRmax) Following Warfarin Alone
Description: INRmax is the maximum INR over the time points after administration of warfarin alone. INR is the ratio of the actual prothrombin time over normal prothrombin time. Geometric Least Squares (LS) mean model was used that was estimated from a mixed-effects model with repeated measures (MMRM) that included treatment as a fixed effect, and participant as a random effect and a random term error.
Time Frame: Period 1 (8 days): Predose on Day 1, up to 96 hours postdose or Period 2 (19 up to 30 days): Predose on Day 15, up to 96 hours post warfarin dose
Population: All enrolled participants who were assigned to a treatment, received at least 1 dose of study treatment and had at least 1 evaluable INRmax warfarin or warfarin/enzastaurin value.
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Groups:
- Warfarin: Period 1 Day 1 (of an 8 day period): 5 milligrams (mg) warfarin administered as a single oral dose. Period included at least a 7-day washout.
Arm/Group | Warfarin | Warfarin + Enzastaurin
Number analyzed (Participants) | 13 | 10
ratio | 1.18 [1.03 to 1.35] | 1.09 [0.95 to 1.26]
Statistical Analysis 1: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Ratio = 0.92, 90% CI 2-sided [0.86 to 1.00] — Ratio of Geometric LS mean

9. Secondary Outcome: Pharmacodynamics: Area Under International Normalised Ratio-time Curve AUC(INR) Following Warfarin Alone
Description: AUC(INR) is the area under INR time curve over the time after administration of warfarin alone. INR is the ratio of actual prothrombin time over normal prothrombin time. Geometric Least Squares (LS) mean model was used that was estimated from a mixed-effects model with repeated measures (MMRM) that included treatment as a fixed effect, and participant as a random effect and a random term error.
Time Frame: as for outcome 8
Population: All enrolled participants who were assigned to a treatment, received at least 1 dose of study treatment and at least 1 evaluable warfarin or warfarin plus enzastaurin AUC(INR) value.
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Warfarin | Warfarin + Enzastaurin
Number analyzed (Participants) | 13 | 9
ratio | 97.24 [93.52 to 101.11] | 95.45 [91.47 to 99.59]
Statistical Analysis 1: Comparison: Warfarin vs Warfarin + Enzastaurin; Test type: Superiority or Other; Ratio = 0.98, 90% CI 2-sided [0.95 to 1.02] — Ratio of Geometric LS mean

10. Secondary Outcome: Pharmacodynamics: Maximum International Normalised Ratio (INRmax) Following Concomitant Administration of Warfarin and Enzastaurin
Description: INRmax is the maximum INR over the time points after administration of warfarin and enzastaurin. INR is the ratio of the actual prothrombin time over normal prothrombin time. Geometric Least Squares (LS) mean model was used that was estimated from a mixed-effects model with repeated measures (MMRM) that included predose measurement of INR in warfarin alone (Period 1) as a covariate, treatment as a fixed effect, participant as a random effect and a random error term. (See Outcome Measure 8 for statistical analysis comparing reporting groups Warfarin and Warfarin co-administered with Enzastaurin)
Time Frame: Period 2 Day 15 (19 up to 30 days): Predose, up to 96 hours post warfarin dose
Population: All enrolled participants who were assigned to a treatment, received at least 1 dose of study treatment and had at least 1 evaluable INRmax warfarin and enzastaurin value.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Groups:
- Warfarin + Enzastaurin: Period 2 (19 up to 30 days): 500 milligrams (mg) enzastaurin administered orally once daily for at least 19 consecutive days and 5 mg warfarin administered as a single oral dose on Day 15.
Arm/Group | Warfarin + Enzastaurin
Number analyzed (Participants) | 10
ratio | 1.09 [0.95 to 1.26]

11. Secondary Outcome: Pharmacodynamics: Area Under International Normalised Ratio-Time Curve AUC(INR) Following Concomitant Administration of Warfarin and Enzastaurin
Description: AUC(INR) is the area under INR time curve over the time after administration of warfarin and enzastaurin. INR is the ratio of actual prothrombin time over normal prothrombin time. Geometric Least Squares (LS) mean model was used that was estimated from a mixed-effects model with repeated measures (MMRM) that included predose measurement of INR in warfarin alone (Period 1) as a covariate, treatment as a fixed effect, participant as a random effect and a random error term. (See Outcome Measure 9 for statistical analysis comparing reporting groups Warfarin and Warfarin co-administered with Enzastaurin.)
Time Frame: Period 2 Day 15 (19 up to 30 days): Predose, up to 96 hours post warfarin dose
Population: All enrolled participants who were assigned to a treatment, received at least 1 dose of study treatment and at least 1 evaluable AUC(INR) concomitant warfarin and enzastaurin value.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | Warfarin + Enzastaurin
Number analyzed (Participants) | 9
ratio | 95.45 [91.47 to 99.59]

12. Secondary Outcome: Pharmacodynamics: International Normalised Ratio (INR) Following Enzastaurin Alone
Description: INR is the ratio of the actual prothrombin time over normal prothrombin time. Geometric Least Squares (LS) mean model was used that was estimated from timepoint (Period 1 Lead-in Day, 0 and 4 hours at Period 2, Day 14) as fixed effect, participant as a random effect and a random error term.
Time Frame: Period 2 Day 14 (19 up to 30 days): Predose and 4 hours postdose
Population: All enrolled participants who were assigned to a treatment, received at least 1 dose of study treatment and at least 1 evaluable INR enzastaurin result.
Measure: Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Enzastaurin
Number analyzed (Participants) | 10
ratio
  Period 2, Day 14, 0 Hours | 0.97 [0.92 to 1.02]
  Period 2, Day 14, 4 Hours | 0.96 [0.91 to 1.01]
Statistical Analysis 1: Comparison: Enzastaurin; Test type: Superiority or Other; Ratio of Geometric LS Mean = 1.03, 90% CI [0.99 to 1.08] — Ratio of Geometric LS mean for Period 2, Day 14, 0 hours
Statistical Analysis 2: Comparison: Enzastaurin; Test type: Superiority or Other; Ratio of Geometric LS Means = 1.02, 90% CI 2-sided [0.98 to 1.06] — Ratio of Geometric LS mean for Period 2, Day 14, 4 hours

ADVERSE EVENTS:
Groups:
- Period 1: Period 1 Day 1 (of an 8-day period): 5 milligrams (mg) warfarin administered as a single oral dose. Period included at least a 7-day washout.
- Period 2, Prior to Warfarin Dose: Period 2 (19 up to 30 days): 500 mg enzastaurin administered orally once daily up to Day 14.
- Period 2, Post Warfarin Dose: Period 2 (19 up to 30 days): 500 mg enzastaurin administered orally once daily for at least 19 consecutive days and 5 mg warfarin administered as a single oral dose on Day 15. Enzastaurin administered up to 30 days total.
- Safety Extension: Safety Extension: Participants were allowed to continue receiving 500 mg enzastaurin orally once daily alone until disease progression or other discontinuation criteria are met.
  Participants were on study for up to a total 8 months (Period 1, Period 2 and Safety Extension).
Arm/Group | Period 1 | Period 2, Prior to Warfarin Dose | Period 2, Post Warfarin Dose | Safety Extension
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 5/13 | 8/12 | 7/10 | 5/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Period 1 (N=13) | Period 2, Prior to Warfarin Dose (N=12) | Period 2, Post Warfarin Dose (N=10) | Safety Extension (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Ocular icterus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iodine allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0/7 (0) | 0/7 (0) | 1/5 (1) | 0/3 (0)
Tooth avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1/7 (1) | 0/7 (0) | 0/5 (0) | 0/3 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1/7 (1) | 0/7 (0) | 0/5 (0) | 0/3 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days